CLINICAL TRIAL: NCT01360684
Title: Pilot Study of Measuring Axillary Skin Temperature, Using DuoFertility, as a Marker of Ovulation in 10 Women of Childbearing Age
Brief Title: Study of Axillary Skin Temperature as a Marker of Ovulation
Status: Completed | Type: Observational
Sponsor: Joanne Outtrim (Other)
Collaborators: Cambridge Temperature Concepts (Industry)
Responsible Party: Sponsor-Investigator, Joanne Outtrim, Senior Research Nurse, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Other Study IDs: A091932; 10/H0308/35 (Other: National Research Ethics Committee)
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Infertility is the most common reason women (aged 20-45yrs)see their GP, affecting 1 in 7 couples. Measuring basal body temperature is a technique that has been used since the 1930's to attempt to predict ovulation. Current NICE guidelines don't recommend the use of BBT charts to predict ovulation, as it has not been established to reliably confirm ovulation.

The DuoFertility sensor a CE marked Class la device provides a continuous accurate measure of axilla temperature whilst worn under the arm.

The investigators plan to compare the temperature measurements of the DuoFertility sensor with the gold standard transvaginal ultrasound scan obtained during 10 infertile women's menstrual cycles, up to 10 cycles per women.

The investigators aim to investigate if continuous axillary skin temperature measurement obtained from the DuoFertility sensor, provides comparable results for identifying the occurrence of ovulation as the gold standard transvaginal ultrasound scan.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation
* Females aged 18 to 44 years.
* Referred with infertility to the Reproductive Medicine Clinic, Rosie Hospital
* Have a body mass index (BMI) above 19 and below 29
* Regular menstrual cycles, i.e. no greater than 7 days difference between the shortest and longest cycle in the last 6 months
* Minimum menstrual cycle 21 days
* Maximum menstrual cycle 35 days
* Willing to wear a DuoFertility sensor continuously for 8 to 10 menstrual cycles;
* Willing to attend Rosie Hospital up to 5 times per cycle for TVS and blood tests
* Willing to perform twice daily LH urine tests at home from day 8 of cycle till positive
* Normal pelvic ultrasound and blood results obtained during screening tests

Exclusion Criteria:

* Aged younger than 18 years, or older than 44 years
* Have a BMI less than 18 or greater than 29
* Any diagnosed systemic illnesses, including but not restricted to thyroid disease, diabetes or inflammatory diseases
* Polycystic ovary disease
* Endometriosis or other pelvic pathology (including proven tubal disease)
* Taking steroids, including oral contraceptives or anti inflammatory drugs

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Infertile females of child bearing age with regular menstrual cycles trying to get pregnant
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raj Mathur, Principal Investigator — Cambridge University Hospital NHS Foundation Trust
Locations (1):
- Cambridge University Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom